CLINICAL TRIAL: NCT00192777
Title: Concurrent Xeloda and Radiotherapy for Bone Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BM-RT-Xeloda.CTIL
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2007-10-08 (Estimated); Status verified 2005-09

CONDITIONS: Solid Tumors; Bone Metastases
Keywords: Solid Tumors; Bone Metastases; Radiotherapy; Xeloda; Concurrent; Radiosensitization
MeSH Terms: interventions — Capecitabine

INTERVENTIONS:
Drug: Xeloda
Procedure: External Beam Radiotherapy

SUMMARY:
Hypothesis: Radiosensitization using Xeloda should improve the rate of complete pain relief.

Primary Objective:

* To determine the frequency of pain relief for the proposed regimen.

Secondary Objective(s):

* To determine the duration of pain relief and narcotic relief for the proposed regimen.
* To determine the frequency of narcotic relief for the proposed regimen.
* To determine the toxicity of concurrent UFT and radiotherapy in patients with bone metastases.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be 18 years of age or older.
2. The patient must have epithelial malignancy.
3. Radiographic evidence of bone metastasis is required. Acceptable studies include plain radiographs, radionuclide bone scans, computed tomography scans and magnetic resonance imaging.
4. The patient must have pain that appears to be related to the radiographically documented metastasis.
5. Patients must have an estimated life expectancy of 3 months or greater.
6. Signed study-specific informed consent.
7. Karnofsky performance status  40.
8. Calculated creatinine clearance > 50 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-11

PRIMARY OUTCOMES:
The frequency of pain relief for the proposed regimen, using a scale that takes into account the subjective feeling and the use of analgesics | after 3 months

SECONDARY OUTCOMES:
The duration of pain relief and narcotic relief for the proposed regimen after one year
The frequency of narcotic relief for the proposed regimen after one year
The toxicity of concurrent UFT and radiotherapy in patients with bone metastases after one year

CONTACTS AND LOCATIONS:
Overall Officials: Kuten Abraham, Prof., Principal Investigator — Dept. of Oncology, Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel